CLINICAL TRIAL: NCT06417047
Title: Effect of Hand Holding on Reducing Intramuscular Injection-Induced Pain and Anxiety: A Randomized Controlled Study
Brief Title: Effect of Hand Holding on Pain and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Serpil SU, Assistant professors, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Necmettin Erbakan U
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Pain and Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor) The patients will be informed about the study and their consent will be obtained without explaining which group they are in. Since the researcher manages the implementation process of the study, researcher blinding cannot be done. In addition, it will be ensured that the researcher learns which group the patients are in after the patients accept to participate in the study. Thus, the internal validity of the research will be ensured.
  At the same time, blind technique will be applied in terms of statistical analysis in the research. The data will be recorded on the computer by the researcher without using the expression of experimental and control groups, and data analysis will be done by another statistician other than the person who made the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hand Holding Group (Experimental): In the experimental group, hand holding will be done by the researcher, and intramuscular injection will be done by the clinical nurse. All intramuscular injections will be performed by a single nurse and the ventrogluteal region will be used as the injection site. Patients will first fill out the Voluntary Information and Consent Form, and then the Descriptive Characteristics Form and State Anxiety Scale. After the injection site is evaluated, the researcher will hold the patient's hand, the nurse will enter the tissue at a 90-degree angle and administer the drug slowly (1 ml/10 seconds). After removing the needle from the tissue, the nurse will apply pressure with dry cotton, and then the researcher will stop holding the patient's hand. After the procedure, the Numerical Pain Scale and State Anxiety Scale will be filled in within 1 minute.
  Interventions: Other: Hand Holding
- Control Group (No Intervention): In the control group, intramuscular injection will be performed by the clinic nurse. All intramuscular injections will be performed by a single nurse and the ventrogluteal region will be used as the injection site. Patients will first fill out the Voluntary Information and Consent Form, and then the Descriptive Characteristics Form and State Anxiety Scale. After the injection site is assessed, the nurse will enter the tissue at a 90-degree angle and administer the medication slowly (1 ml/10 seconds). After removing the needle from the tissue, the nurse will apply pressure with dry cotton. After the procedure, the Numerical Pain Scale and State Anxiety Scale will be filled in within 1 minute.

INTERVENTIONS:
Other: Hand Holding — During the intramuscular injection, the aim is to draw the patients' attention elsewhere by holding their hand.
  Arms: Hand Holding Group

SUMMARY:
It was aimed to examine the effect of the hand holding method applied during intramuscular injection on pain and anxiety.

DETAILED DESCRIPTION:
This study was designed as a pre-test-post-test regular parallel group, randomized controlled experimental design. The research will be carried out in the Adult Emergency Service of the Ministry of Health of the Republic of Turkey, Konya City Hospital. Patients will be randomly divided into two groups: handholding (52) and control group (52). For the Hand Holding Group: After the patient is positioned appropriately, the patient's hand will be held by the researcher. Once the intramuscular injection is completed, the patient's hand holding will be stopped. For the Control Group: No application will be made during intramuscular injection in the control group. The primary outcome of this study is to determine patients' pain scores during the intramuscular injection procedure. The secondary outcome is to determine the anxiety levels of patients.

ELIGIBILITY:
Inclusion Criteria:

* Having vitamin B 12 1000 mcg/ml (1 ml ampoule) intramuscular treatment,
* Being literate,
* Are between the ages of 18-65,
* No visual, hearing, sensory or motor loss or cognitive impairment,
* Not using centrally or peripherally acting analgesics or sedatives,
* There is no scar tissue, incision, lipodystrophy or signs of infection on the skin of the injection area,
* Having a body mass index between 18.5 and 29.5,
* Injected into the ventrogluteal area,
* Individuals who agree to participate in the research will be included.

Exclusion Criteria:

* Those with chronic pain,
* Having a psychiatric disorder,
* Foreign nationals,
* Patients with contact-communicable diseases will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2024-07-20 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Scale | It will be filled within 1 minute after the intramuscular injection is completed.
  A score of "0" indicated the lowest pain, and a score of "10" indicated the highest pain.

SECONDARY OUTCOMES:
State Anxiety Scale | It will be filled immediately before the intramuscular injection and within 1 minute after the procedure is completed.
  A score between 20-80 is obtained. The highest score obtained from the scale indicates a high level of anxiety, while a low score indicates a low level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Serpil SU, Study Chair — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No